CLINICAL TRIAL: NCT00044525
Title: An Uncontrolled Phase II Study Evaluating the Efficacy and Safety of Intravenous BAY59-8862 in Patients With Taxane-Resistant Metastatic Breast Cancer
Brief Title: Evaluation of BAY59-8862 in Taxane-Resistant Metastatic Breast Cancer Patients
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 10654
Record Dates: First submitted 2002-08-30; First posted 2002-09-04 (Estimated); Last update posted 2014-12-23 (Estimated); Status verified 2014-12

CONDITIONS: Breast Neoplasms; Breast Cancer, Metastatic
Keywords: Taxane; Breast Cancer; Metastasis
MeSH Terms: conditions — Breast Neoplasms; Neoplasm Metastasis | interventions — IDN 5109

ARMS (1):
- Arm 1 (Experimental)
  Interventions: Drug: BAY59-8862 (Cytotoxic Taxane)

INTERVENTIONS:
Drug: BAY59-8862 (Cytotoxic Taxane) — 1 h intravenous infusion every 3 weeks

SUMMARY:
Breast cancer is the most common form of cancer among women in developing countries, accounting for approximately one-fifth of all female cancers in the United States. Although mortality rates are declining in some countries, it remains the leading cause of death in women aged 40-55 years. The median survival for women with metastatic breast cancer is 2-3 years but there is significant variability in this population. The primary goals of treatment in patients with metastatic breast cancer are improvement or maintenance of quality of life and prolongation of survival. The taxanes, paclitaxel and docetaxel, were incorporated into the treatment of metastatic breast cancer in the 1990's. The usefulness of the taxanes is limited by the development of tumor resistance to these agents. This phase II trial with BAY59-8862 will be conducted to determine the anti-tumor efficacy of BAY59-8862 in taxane-resistant metastatic breast cancer.

ELIGIBILITY:
Inclusion Criteria:

* Female patients with a proven diagnosis of metastatic breast cancer
* Measurable disease as defined by the presence of at least one measurable lesion
* Patients must have received at least 3 weeks of continuous therapy with Taxane
* patient must subsequently develop progressive disease either during treatment or within 6 months after treatment
* Patients who failed on hormone therapy
* Life expectancy of at least 12 weeks.
* Adequate bone marrow, liver and kidney function
* Patients with active brain metastases may be included

Exclusion Criteria:

* Excluded medical conditions like: pre-existing neuropathy, active heart diseases or ischemia; surgery within 4 weeks of study entry; serious infections; HIV infection; chronic hepatitis B or C; patients with brain metastases must be without a seizure; hypersensitivity to taxanes; organ transplants; some previous cancers
* Excluded therapies and medications, previous and concomitant such as: anticancer chemotherapy or immunotherapy during the study or within 4 weeks prior to study entry; more than two prior anticancer chemotherapy regimens; radiotherapy during study or within 4 weeks prior to study entry; bone marrow transplant
* Others: pregnant or breast-feeding patients; women enrolled in this trial must use adequate barrier birth control measures during the course of the trial; substance abuse, medical, psychological or social conditions that may interfere with the patient's participation.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 82 (Actual)
Dates: Start 2002-04; Primary Completion 2004-02 (Actual); Study Completion 2004-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (20):
- Germany (3):
  - Stuttgart, Baden-Wurttemberg
  - Berlin, State of Berlin
  - Jena, Thuringia
- Greece (2):
  - Marousi, Attica
  - Heraklion, Crete
- Israel (4):
  - Ashkelon
  - Haifa
  - Tel Aviv
  - Tel Litwinsky
- Italy (7):
  - Treviglio, Bergamo
  - Rozzano, Milano
  - Biella
  - Cuneo
  - Forlì
  - Parma
  - Udine
- Poland (2):
  - Olsztyn
  - Warsaw
- Aarau, Canton of Aargau, Switzerland
- London, Greater London, United Kingdom